CLINICAL TRIAL: NCT05311280
Title: The Effect of High Intensity Interval Exercise and Myofunctional Therapy on Obstructive Sleep Apnea: a Randomized Clinical Controlled Trial
Brief Title: The Effect of High Intensity Interval Exercise and Myofunctional Therapy on Obstructive Sleep Apnea
Acronym: OSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYGH109058
Record Dates: First submitted 2021-10-04; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Myotherapy; High intensity interval training
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: intervention group: Myotherapy+High intensity interval training Control group: Myotherapy + general home exercise
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intensity interval training plus myotherapy (Experimental): Subjects were instructed to perform tongue slide, tongue force, tongue press, tongue reach, swallowing exercise, smiling exercise, jaw press exercise, chewing exercise, breathing exercise and buccinator exercise.These myofunctional exercise were performed 10 repetitions for a set, 2 sets in a treatment session depends on patient's condition. Between each session, subjects were allowed to rest at least 1 minutes.
  Exercise training would be implemented in the form of high-intensity interval training and resistance exercise. High-intensity interval training intensity of the target heart rate (THR) was calculated as follows: THR = (HRmax - HRrest) × 80-90%Intensity + HRrest[26]. The HIIT program included four 3-min bouts at high-intensity (80-90%HRR), separated by 3-min of active recovery and total for 4 cycles of 24-min HIIT intervention. The HIIT exercise options were running on a treadmill.
  Interventions: Other: high intensity interval training plus myotherapy
- home exercise training plus myotherapy (Active Comparator): Subjects were instructed to perform tongue slide, tongue force, tongue press, tongue reach, swallowing exercise, smiling exercise, jaw press exercise, chewing exercise, breathing exercise and buccinator exercise.These myofunctional exercise were performed 10 repetitions for a set, 2 sets in a treatment session depends on patient's condition.
  Home exercise is composed of ambulation training outside or inside. Three phase including warm up, training phase, and cool down. The intensity of training phase is decided by rating of perceived exertion (RPE) range from 11~15. 2~5 training times a week will involved according to patients' preference.
  Interventions: Other: home exercise plus myotherapy

INTERVENTIONS:
Other: high intensity interval training plus myotherapy — High intensity interval training (HIIT) has been proved its same effect on lower down body fat as moderate intensity continuous training (MICT). In addition, HIIT has the additional benefit of being a time-efficient program which can increase exercise adherence and the participants were more likely to intend to continue. Previous two studies show that HIIT could improve the severity of OSA in both obese adults and obese children.
  Myotherapy: MT is composed of isotonic and isometric exercise related to oral, oropharyngeal, and respiratory exercise. Based on previous review and meta-analysis, MT can decrease not only AHI score, but also ESS score. It means that MT is beneficial to release the symptom of sudden apnea and hypopneas.
  Arms: high intensity interval training plus myotherapy
Other: home exercise plus myotherapy — Home exercise: ambulation by patients themselves Myotherapy: MT is composed of isotonic and isometric exercise related to oral, oropharyngeal, and respiratory exercise. Based on previous review and meta-analysis, MT can decrease not only AHI score, but also ESS score. It means that MT is beneficial to release the symptom of sudden apnea and hypopneas.
  Arms: home exercise training plus myotherapy

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep disorder which is caused because of collapse of airway or inappropriate tongue position. As OSA becomes severe, the physical and psychological aspect might be influenced due to insomnia. In addition, many evidences revealed that OSA is related to cardiovascular disorder. Apnea-hypopnea index (AHI) and epworth sleepiness scale (ESS) are common parameters to evaluate the severity of OSA. Recently, body and tongue fat have certain relation with OSA, and the higher the fat, the more possible to get OSA. To find the treatments for OSA, myotherapy has been proved to improve AHI and ESS. The treat mechanism is speculated that increasing muscle tone around oral and oropharyngeal and decreasing tongue fat. High intensity interval training (HIIT) might be effective to OSA, for it could lower down the total body fat. Furthermore, HIIT is a time-efficient program which can increase exercise adherence. Last, less articles discussed about the effect of supervised verse unsupervised treatment and the effect of mix-model treatment. The purpose of the study is investigating the comparison between supervised HIIT plus myotherapy and unsupervised home exercise plus myotherapy.

Method:

40 patients who meets the inclusion criteria will be recruited in this article during 2022/01 to 2022/12. Then, they will be randomly assigned into HIIT plus myotherapy group and home exercise plus myotherapy group. The treatment process will last for 8 weeks. All the outcomes such as AHI,ESS and body fat will be completed before and after 8 weeks treatment. The Wilcox signed test was adopted to analyze the treatment before and after the treatment sessions (time effect). The Mann-Whitney U was applied for the difference before and after treatment between two groups (group effect), and the baseline of two groups was also analyzed by this method. The significant level was set as p value< 0.05.

Hypothesis:

It is speculated that HIIT plus myotherapy might revealed better outcomes on AHI, ESS, and body fat.

DETAILED DESCRIPTION:
1. introduction Obstructive sleep apnea (OSA) is a sleep disorder that is characterized by apneas and hypopneas during sleep due to repetitive collapse of the upper airway. The prevalence is 3-7% in men and 2-5% in women. Daytime sleepiness and insomnia are associated with both decreased physical activity and increased obesity, increased OSA severity is also associated with decreased physical activity, resulting in a vicious cycle. Accumulating evidence shows that OSA is associated with multiple cardiovascular disorders, such as hypertension, type 2 diabetes mellitus and coronary artery disease. The treatment of OSA may reduce the risk of these cardiovascular disorders. The apnea-hypopnea index (AHI) has been widely used to quantify the level of OSA by the number of apnea episodes per hour. Based on the definition of American Academy of Sleep Medicine (AASM) and an article about epidemiology of OSA, AHI range from 5~15 is defined as mild OSA, and AHI 15~30 is defined as moderate OSA. AHI over 30 can be regarded as severe OSA. Epworth sleepiness scale (ESS) is a questionnaire to measure subject general level of daytime sleepiness. OSA patients often revealed higher score which refers to higher possibility to get sleep disorder. Recently, some articles showed that body and tongue fat deposition have certain relation with OSA, the higher the fat, the more possible to get OSA. Body fat can be quantified through waist and neck circumference.

   In order to solve OSA, myotherapy (MT) might be an effective method. MT is composed of isotonic and isometric exercise related to oral, oropharyngeal, and respiratory exercise. Based on previous review and meta-analysis, MT can decrease not only AHI score, but also ESS score. It means that MT is beneficial to release the symptom of sudden apnea and hypopneas through decreasing the amount of fatty deposition of the tongue and increasing oral and oropharyngeal muscle tone. Recent article also supports that weight and fat loss of soft tissue of tongue is important for treat OSA[12]. Some articles also mentioned that the snoring situation during sleep time has declined. That is, the sleep interruption to people sleeping beside the OSA patient are alleviated. In addition, the sleep and life quality can be ameliorated by myotherapy. Inconsistent evidence also manifested that oxygen saturation has been improved after myotherapy. In short, MT can be regarded as optimal alternative therapy to mild to moderate OSA patient.

   Exercise training is an effective intervention in reducing the severity of OSA and improving symptoms of sleepiness and quality of life. According to previous systematic review and meta-analysis, exercise such as aerobic exercise and resistance exercise has been proved effective on improving AHI, ESS. However, these articles didn't focus on body fat that is highly associated with OSA. According to recent article, decreasing body fat is essential to deal with OSA. Hence, high intensity interval training (HIIT) has been proved its same effect on lower down body fat as moderate intensity continuous training (MICT). HIIT also shows greater effectiveness compared with (MICT) on cardiovascular and metabolic function in both healthy populations and populations with cardiovascular disease. In addition, HIIT has the additional benefit of being a time-efficient program which can increase exercise adherence and the participants were more likely to intend to continue. Previous two studies show that HIIT could improve the severity of OSA in both obese adults and obese children, but it still needs evidence to prove the effectiveness among different aspects.

   According to recent literature review, there is no standard physical therapy model for OSA. Furthermore, less articles discussed about the effect of supervised verse unsupervised treatment and the effect of mix-model treatment. Hence, the purpose of the study is investigating the comparison between supervised HIIT plus myotherapy and unsupervised home exercise plus myotherapy. It is hypothesized that HIIT plus myotherapy might revealed better outcomes on AHI, ESS, and body fat.
2. Method Procedure The subjects included in this study were randomized assigned to experimental group and control group. The randomization orders were decided by computer, and all the contents were concealed into a dark color envelop. Before first treatment, the envelops were opened to determine which treatment protocol were adopted. The treatment of experimental group was composed of myotherapy and resistance exercise plus high intensity interval training (HIIT). The treatment of control group was composed of general stretch exercise plus myotherapy. Subsequently, initial measurement was conducted including BMI, Body fat, waist and neck circumstanced, apnea hypopnea index (AHI), Epworth Sleepiness Scale (ESS), oxygen desaturation index (ODI) and body fat. Then, the treatment protocols were both executed for 30 minutes, sixteen times in two months. After completing the treatment process, the final measurement was conducted as the initial treatment. All the outcomes were collected and analyzed by statistically method.

Treatment Experimental group is composed of myotherapy and high intensity interval training (HIIT) plus resistance exercise. Myotherapy was based on the studies by Lequeux et al. and Cláudia et al. Subjects were instructed to perform tongue slide, tongue force, tongue press, tongue reach, swallowing exercise, smiling exercise, jaw press exercise, chewing exercise, breathing exercise and buccinator exercise. Exercise training would be implemented in the form of high-intensity interval training and resistance exercise. High-intensity interval training intensity of the target heart rate (THR) was calculated as follows: THR = (HRmax - HRrest) × 80-90%Intensity + HRrest. The HIIT program included four 3-min bouts at high-intensity (80-90%HRR), separated by 3-min of active recovery and total for 4 cycles of 24-min HIIT intervention. The HIIT exercise options were running on a treadmill. Polar heart rate monitors were used to monitor exercise intensity. Subsequently, the 20-min resistance exercise program was conducted using a theraband. The different colors of band indicate different levels of resistance. The four limbs were mainly exercised with yellow, red, green and blue colored elastic bands. In this regard, the theraband was color-coded in the following order of increasing resistance: blue, green, blue and dark. Each subject began the program using the blue theraband. As the subjects performed the ability to complete 15 repetitions without difficulty, the intensity of the thraband was progressed. The volume of the resistance was 10 repetitions per set, and 3 set in a training session. Exercises included shoulder press, shoulder lateral raise, biceps curl, butterfly, seat row, leg press(squat), calf raise, latissmus pulldown, abdominal curl and bridge. Five minutes of stretching exercises was conducted as a warm-up and cool down period before and after training sessions. The physiotherapist with abundant experience related to myotherapy and high intensity interval training (HIIT) plus resistance exercise supervised all the treatment process to confirm the quality of execution. This exercise was performed 12~15 repetition depends on patient's condition.

Statistical analysis The primary variable of the study were body fat, neck and waist circumstance, AHI, ODI and ESS. The secondary variable of the study were body weight and BMI. Descriptive statistics for the categorical variable were documented as frequency counts and percentages. The continuous variables were reported as mean + SD, if they were normal distribution, or they were recorded as median and range.

The Wilcox signed test was adopted to analyze the treatment before and after the treatment sessions (time effect). The Mann-Whitney U was applied for the difference before and after treatment between two groups (group effect), and the baseline of two groups was also analyzed by this method. The significant level was set as p value< 0.05. All the statistical data analysis was performed by SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis as OSA by ENT
* AHI 5~30 (mild to moderate OSA)
* BMI >24
* Body fat male>20% female>30%
* age from 20~80

Exclusion Criteria:

* Rest BP < 160/100
* Unstable cardiopulmonary disease
* CPAP use
* mandibular advancement
* Cancer
* BMI > 40
* unable to speak Chinese or English

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | Change from baseline Apnea-hypopnea index for 2 month
  The severity of sleep apnea was evaluated by an apnea-hypopnea index (AHI; number of apneas and hypopneas per hour of sleep) according to the data of polysomnography (PSG) in sleep center of TYGH. The average number of desaturation episodes per hour
Epworth Sleepiness Scale (ESS) | Change from baseline Epworth Sleepiness Scale for 2 month
  The excessive daytime sleepiness was measured by Epworth Sleepiness Scale (ESS)
body fat | Change from baseline body fat for 2 month
  Total body fat was evaluated by the weight scale that is correction by Inbody machine with high validity
waist and neck circumstance | change from baseline waist and neck circumstance for 2 month
  he waist and neck circumstance were measured by measuring tape

SECONDARY OUTCOMES:
oxygen desaturation index (ODI) | change from baseline oxygen desaturation index for 2 month
  The ODI is measured by an oximeter, which is a device typically placed on the fingertip that shines a red light on the skin and can estimate the amount of oxygen in the peripheral blood. Desaturation episodes are generally described as a decrease in the mean oxygen saturation of ≥4% (over the last 120 seconds) that lasts for at least 10 seconds. The ODI was graded into three groups: mild (5-14), moderate (15-29), and severe (≥30) OSA. Patients with an ODI<5 were graded as having no oxygen disturbance
BMI | change from baseline BMI for 2 month
  Total body fat was evaluated by the weight scale that is correction by Inbody machine with high validity. The parameters such as BMI and body fat mass were measured by this test.

CONTACTS AND LOCATIONS:
Locations (1):
- Taoyaun General Hospital, Ministry of Wealth and Health, Taoyuan District, Taoyuan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Background] Franklin KA, Lindberg E. Obstructive sleep apnea is a common disorder in the population-a review on the epidemiology of sleep apnea. J Thorac Dis. 2015 Aug;7(8):1311-22. doi: 10.3978/j.issn.2072-1439.2015.06.11. PMID 26380759
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Chasens ER, Sereika SM, Weaver TE, Umlauf MG. Daytime sleepiness, exercise, and physical function in older adults. J Sleep Res. 2007 Mar;16(1):60-5. doi: 10.1111/j.1365-2869.2007.00576.x. PMID 17309764
- [Background] Chasens ER, Sereika SM, Houze MP, Strollo PJ. Subjective and objective appraisal of activity in adults with obstructive sleep apnea. J Aging Res. 2011 Jan 3;2011:751819. doi: 10.4061/2011/751819. PMID 21253491
- [Background] Quan SF, O'Connor GT, Quan JS, Redline S, Resnick HE, Shahar E, Siscovick D, Sherrill DL. Association of physical activity with sleep-disordered breathing. Sleep Breath. 2007 Sep;11(3):149-57. doi: 10.1007/s11325-006-0095-5. PMID 17221274
- [Background] Tietjens JR, Claman D, Kezirian EJ, De Marco T, Mirzayan A, Sadroonri B, Goldberg AN, Long C, Gerstenfeld EP, Yeghiazarians Y. Obstructive Sleep Apnea in Cardiovascular Disease: A Review of the Literature and Proposed Multidisciplinary Clinical Management Strategy. J Am Heart Assoc. 2019 Jan 8;8(1):e010440. doi: 10.1161/JAHA.118.010440. No abstract available. PMID 30590966
- [Background] Yacoub M, Youssef I, Salifu MO, McFarlane SI. Cardiovascular Disease Risk in Obstructive Sleep apnea: An Update. J Sleep Disord Ther. 2017;7(1):283. doi: 10.4172/2167-0277.1000283. Epub 2018 Feb 12. No abstract available. PMID 29644149
- [Background] Gilat H, Vinker S, Buda I, Soudry E, Shani M, Bachar G. Obstructive sleep apnea and cardiovascular comorbidities: a large epidemiologic study. Medicine (Baltimore). 2014 Aug;93(9):e45. doi: 10.1097/MD.0000000000000045. PMID 25144324
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Kim AM, Keenan BT, Jackson N, Chan EL, Staley B, Poptani H, Torigian DA, Pack AI, Schwab RJ. Tongue fat and its relationship to obstructive sleep apnea. Sleep. 2014 Oct 1;37(10):1639-48. doi: 10.5665/sleep.4072. PMID 25197815
- [Background] Wang SH, Keenan BT, Wiemken A, Zang Y, Staley B, Sarwer DB, Torigian DA, Williams N, Pack AI, Schwab RJ. Effect of Weight Loss on Upper Airway Anatomy and the Apnea-Hypopnea Index. The Importance of Tongue Fat. Am J Respir Crit Care Med. 2020 Mar 15;201(6):718-727. doi: 10.1164/rccm.201903-0692OC. PMID 31918559
- [Background] Iftikhar IH, Kline CE, Youngstedt SD. Effects of exercise training on sleep apnea: a meta-analysis. Lung. 2014 Feb;192(1):175-84. doi: 10.1007/s00408-013-9511-3. PMID 24077936
- [Background] Bollens B, Reychler G. Efficacy of exercise as a treatment for Obstructive Sleep Apnea Syndrome: A systematic review. Complement Ther Med. 2018 Dec;41:208-214. doi: 10.1016/j.ctim.2018.10.002. Epub 2018 Oct 3. PMID 30477841
- [Background] Aiello KD, Caughey WG, Nelluri B, Sharma A, Mookadam F, Mookadam M. Effect of exercise training on sleep apnea: A systematic review and meta-analysis. Respir Med. 2016 Jul;116:85-92. doi: 10.1016/j.rmed.2016.05.015. Epub 2016 May 21. PMID 27296826
- [Background] Fisher G, Brown AW, Bohan Brown MM, Alcorn A, Noles C, Winwood L, Resuehr H, George B, Jeansonne MM, Allison DB. High Intensity Interval- vs Moderate Intensity- Training for Improving Cardiometabolic Health in Overweight or Obese Males: A Randomized Controlled Trial. PLoS One. 2015 Oct 21;10(10):e0138853. doi: 10.1371/journal.pone.0138853. eCollection 2015. PMID 26489022
- [Background] Jelleyman C, Yates T, O'Donovan G, Gray LJ, King JA, Khunti K, Davies MJ. The effects of high-intensity interval training on glucose regulation and insulin resistance: a meta-analysis. Obes Rev. 2015 Nov;16(11):942-61. doi: 10.1111/obr.12317. PMID 26481101
- [Background] Heinrich KM, Patel PM, O'Neal JL, Heinrich BS. High-intensity compared to moderate-intensity training for exercise initiation, enjoyment, adherence, and intentions: an intervention study. BMC Public Health. 2014 Aug 3;14:789. doi: 10.1186/1471-2458-14-789. PMID 25086646
- [Background] Karlsen T, Nes BM, Tjonna AE, Engstrom M, Stoylen A, Steinshamn S. High-intensity interval training improves obstructive sleep apnoea. BMJ Open Sport Exerc Med. 2017 Feb 8;2(1):bmjsem-2016-000155. doi: 10.1136/bmjsem-2016-000155. eCollection 2016. PMID 29616142
- [Background] Longlalerng K, Sonsuwan N, Uthaikhup S, Kietwatanachareon S, Kamsaiyai W, Panyasak D, Pratanaphon S. High-intensity interval training combined with resistance training improved apnea-hypopnea index but did not modify oxygen desaturation index and oxygen saturation nadir in obese children with obstructive sleep apnea. Sleep Breath. 2020 Jun;24(2):571-580. doi: 10.1007/s11325-019-01899-z. Epub 2019 Jul 23. PMID 31338769
- [Background] Emami E, Heydecke G, Rompre PH, de Grandmont P, Feine JS. Impact of implant support for mandibular dentures on satisfaction, oral and general health-related quality of life: a meta-analysis of randomized-controlled trials. Clin Oral Implants Res. 2009 Jun;20(6):533-44. doi: 10.1111/j.1600-0501.2008.01693.x. PMID 19515032
- [Background] Patel S, Kon SSC, Nolan CM, Barker RE, Simonds AK, Morrell MJ, Man WD. The Epworth Sleepiness Scale: Minimum Clinically Important Difference in Obstructive Sleep Apnea. Am J Respir Crit Care Med. 2018 Apr 1;197(7):961-963. doi: 10.1164/rccm.201704-0672LE. No abstract available. PMID 28961021
- [Background] Lequeux T, Chantrain G, Bonnand M, Chelle AJ, Thill MP. Physiotherapy in obstructive sleep apnea syndrome: preliminary results. Eur Arch Otorhinolaryngol. 2005 Jun;262(6):501-3. doi: 10.1007/s00405-004-0806-0. Epub 2004 Dec 30. PMID 15625609
- [Background] de Felicio CM, da Silva Dias FV, Trawitzki LVV. Obstructive sleep apnea: focus on myofunctional therapy. Nat Sci Sleep. 2018 Sep 6;10:271-286. doi: 10.2147/NSS.S141132. eCollection 2018. PMID 30233265
- [Background] Karl G. Stoedefalke, o.A.F., Anne R. Abbott,, The 10th edition of ACSM's Guidelines for Exercise Testing and Prescription. 2018(Exercise Prescription for Patients with Cardiac, Peripheral, Cerebrovascular, and Pulmonary Disease).